CLINICAL TRIAL: NCT00000160
Title: Diabetic Retinopathy Study (DRS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-62
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-06-02 (Estimated); Status verified 2003-10

CONDITIONS: Diabetic Retinopathy; Blindness
Keywords: Vision Loss
MeSH Terms: conditions — Diabetic Retinopathy; Blindness; Vision Disorders | interventions — Light Coagulation

INTERVENTIONS:
Procedure: Xenon Photocoagulation
Procedure: Argon Photocoagulation
Procedure: Photocoagulation

SUMMARY:
To determine whether photocoagulation helps prevent severe visual loss from proliferative diabetic retinopathy.

To determine whether a difference exists in the efficacy and safety of argon versus xenon photocoagulation for proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
By the 1950s, diabetic retinopathy had become a leading cause of blindness and visual disability in the United States. The use of photocoagulation to treat proliferative retinopathy gained widespread use in ophthalmic practice following its introduction in 1959. However, only a few studies of photocoagulation incorporated any of the basic principles of controlled clinical trials, and these involved inadequate numbers of patients. Consequently, there has been inadequate evidence of the actual value of the procedure. Because of the clinical importance of diabetic retinopathy and the increasing use of photocoagulation in its management, the Diabetic Retinopathy Study (DRS) was begun in 1971. This randomized, controlled clinical trial involved more than 1,700 patients enrolled at 15 medical centers.

One eye of each patient was randomly assigned to immediate photocoagulation and the other to followup without treatment, regardless of the course followed by either eye. The eye chosen for photocoagulation was randomly assigned to either of two treatment techniques, one using an argon laser and the other a xenon arc photocoagulator. Patients were followed at 4-month intervals according to a protocol that provided for measurement of best corrected visual acuity.

Treatment was usually completed in one or two sittings and included scatter (panretinal) photocoagulation extending to or beyond the vortex vein ampulae. The argon treatment technique specified 800 to 1,600, 500-micron scatter burns of 0.1 second duration and direct treatment of new vessels whether on or within one disc diameter of the optic disc (NVD) or outside this area (NVE). Focal treatment was also applied to microaneurysms or other lesions thought to be causing macular edema. Followup treatment was applied as needed at 4-month intervals. The xenon technique was similar, but scatter burns were fewer in number, generally of longer duration, and stronger, and direct treatment was applied only to NVE on the surface of the retina.

ELIGIBILITY:
Patients were eligible if they had best corrected visual acuity of 20/100 or better in each eye and the presence of proliferative diabetic retinopathy in at least one eye or severe nonproliferative retinopathy in both eyes. They could not have had prior treatment with photocoagulation or pituitary ablation, and both eyes had to be suitable for photocoagulation. All eligible patients were younger than 70 years, and the examining physician assessed the outlook for survival and availability for 5 years of followup to be good.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1972-01

REFERENCES:
- [Background] Diabetic retinopathy study. Report Number 6. Design, methods, and baseline results. Report Number 7. A modification of the Airlie House classification of diabetic retinopathy. Prepared by the Diabetic Retinopathy. Invest Ophthalmol Vis Sci. 1981 Jul;21(1 Pt 2):1-226. No abstract available. PMID 7195893
- [Background] Four risk factors for severe visual loss in diabetic retinopathy. The third report from the Diabetic Retinopathy Study. The Diabetic Retinopathy Study Research Group. Arch Ophthalmol. 1979 Apr;97(4):654-5. doi: 10.1001/archopht.1979.01020010310003. PMID 426679
- [Background] The Diabetic Retinopathy Study Research Group; Photocoagulation treatment of proliferative diabetic retinopathy: A short report of long range results., Diabetic Retinopathy Study (DRS) Report Number 4. Proceedings of the 10th Congress of the International Diabetes Federation 1979
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy: relationship of adverse treatment effects to retinopathy severity. Diabetic retinopathy study report no. 5. Dev Ophthalmol. 1981;2:248-61. PMID 7262408
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Ederer F, Podgor MJ. Assessing possible late treatment effects in stopping a clinical trial early: a case study. Diabetic Retinopathy Study report No. 9. Control Clin Trials. 1984 Dec;5(4):373-81. doi: 10.1016/s0197-2456(84)80016-1. PMID 6394209
- [Background] Rand LI, Prud'homme GJ, Ederer F, Canner PL. Factors influencing the development of visual loss in advanced diabetic retinopathy. Diabetic Retinopathy Study (DRS) Report No. 10. Invest Ophthalmol Vis Sci. 1985 Jul;26(7):983-91. PMID 2409053
- [Background] Preliminary report on effects of photocoagulation therapy. The Diabetic Retinopathy Study Research Group. Am J Ophthalmol. 1976 Apr;81(4):383-96. doi: 10.1016/0002-9394(76)90292-0. PMID 944535
- [Background] Ferris FL 3rd, Podgor MJ, Davis MD. Macular edema in Diabetic Retinopathy Study patients. Diabetic Retinopathy Study Report Number 12. Ophthalmology. 1987 Jul;94(7):754-60. doi: 10.1016/s0161-6420(87)33526-2. PMID 3658347
- [Background] Kaufman SC, Ferris FL 3rd, Swartz M. Intraocular pressure following panretinal photocoagulation for diabetic retinopathy. Diabetic Retinopathy Report No. 11. Arch Ophthalmol. 1987 Jun;105(6):807-9. doi: 10.1001/archopht.1987.01060060093040. PMID 3555429
- [Background] Kaufman SC, Ferris FL 3rd, Seigel DG, Davis MD, DeMets DL. Factors associated with visual outcome after photocoagulation for diabetic retinopathy. Diabetic Retinopathy Study Report #13. Invest Ophthalmol Vis Sci. 1989 Jan;30(1):23-8. PMID 2912911
- [Background] Indications for photocoagulation treatment of diabetic retinopathy: Diabetic Retinopathy Study Report no. 14. The Diabetic Retinopathy Study Research Group. Int Ophthalmol Clin. 1987 Winter;27(4):239-53. doi: 10.1097/00004397-198702740-00004. No abstract available. PMID 2447027
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy: the second report of diabetic retinopathy study findings. Ophthalmology. 1978 Jan;85(1):82-106. doi: 10.1016/s0161-6420(78)35693-1. PMID 345173